CLINICAL TRIAL: NCT01450813
Title: The Effect of Rocuronium on the Response of Composite Variability Index (CVI) to Laryngoscopy
Brief Title: The Effect of Neuromuscular Blockade on the Composite Variability Index (CVI) During Laryngoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: COVMOPR0176
Record Dates: First submitted 2011-09-22; First posted 2011-10-12 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Anesthesia; Neuromuscular Blockade
MeSH Terms: interventions — Sodium Chloride; Saline Solution; Rocuronium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (Sham Comparator): Saline 0.06 ml/kg
  Interventions: Drug: Saline 0.06 ml/kg
- Group 2 (Active Comparator): Rocuronium 0.2 mg/kg
  Interventions: Drug: Rocuronium 0.2 mg/kg
- Group 3 (Active Comparator): Rocuronium 0.4 mg/kg
  Interventions: Drug: Rocuronium 0.4 mg/kg
- Group 4 (Active Comparator): Rocuronium 0.6 mg/kg
  Interventions: Drug: Rocuronium 0.6 mg/kg

INTERVENTIONS:
Drug: Saline 0.06 ml/kg — IV Infusion x1 prior to laryngoscopy
  Other Names: Normal Saline
  Arms: Group 1
Drug: Rocuronium 0.2 mg/kg — IV Infusion x1 prior to laryngoscopy
  Other Names: Rocuronium bromide: Zemuron
  Arms: Group 2
Drug: Rocuronium 0.4 mg/kg — IV Infusion x1 prior to laryngoscopy
  Other Names: Rocuronium bromide: Zemuron
  Arms: Group 3
Drug: Rocuronium 0.6 mg/kg — IV Infusion x1 prior to laryngoscopy
  Other Names: Rocuronium bromide: Zemuron
  Arms: Group 4

SUMMARY:
The Bispectral Index (BIS) monitor is used in many operating rooms to provide information to the anesthesiologist about a patient's level of consciousness. The Composite Variability Index (CVI) is a new index that may provide the anesthesiologist with more information about the condition of the patient. The CVI is a measure of the combined variability in BIS (bispectral index) and frontal electromyography (EMG) activity that may be useful in assessing the nociception/anti-nociception balance for patients under general anesthesia.The purpose of this study is to determine if a commonly used anesthetic drug (rocuronium) affects the CVI measurement differently with different doses. Rocuronium is a neuromuscular blocking agent (NMBA) routinely used during surgery. It is expected that the group given the highest dose of rocuronium will have diminished CVI values.

This study will randomize patients to one of four doses of rocuronium: no rocuronium, 0.2, 0.4, and 0.6 milligrams per kilo of body weight; the last dose is the standard amount for adults. It is expected that the group given the highest dose of rocuronium will have diminished CVI values. By including intermediate doses, information about the function of CVI in states of less than full muscle relaxation, or paralysis, will be obtained. This information is critically important for the development of the composite variability index, because during general anesthesia patients are usually maintained in a state of less than full paralysis. If the CVI response to stimulation in the intermediate groups is similar to the group receiving no rocuronium, the monitor may find wide clinical applicability. If the response is similar to the maximal rocuronium group, the index may only be reliable in states with no muscle relaxant, which will greatly limit clinical utility.

DETAILED DESCRIPTION:
Consented subjects randomized to one of four doses of rocuronium will be transported to the operating room and be connected to routine monitors that included a BIS (Covidien), M-Entropy sensor (GE Healthcare) and TOF (train of four) monitor. Following preoxygenation, general anesthesia will be induced with propofol and remifentanil using traditional syringe pumps. The induction doses given and subsequent infusion rates will be determined by utilizing pharmacokinetic (Pk) models (Marsh model for propofol, Minto model for remifentanil). Unconsciousness will be confirmed by performing the usual clinical assessments and by obtaining a BIS value between 40 and 50. Once the subject is unconsciousness, they will be given the assigned dose of rocuronium, after which the study anesthesiologist will perform a laryngoscopy. The anesthesiologist performing the laryngoscopy will not know what dose of rocuronium the subject received. Neuromuscular blockade (NMB) will be monitored by a train-of-four twitch monitor (TOF Watch-SX) at the adductor pollicis muscle (2 HZ, 50mAmp) every 15 seconds.

At three minutes after the rocuronium administration, a standardized 20-second laryngoscopy will be applied. The CVI, entropy, and hemodynamic responses (heart rate, blood pressure measurement each minute) and train-of-four measurements will be monitored for three minutes before and after the laryngoscopy.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesia (ASA) physical status class I or II.
* Body mass index between 18 and 35 kg m-2.
* No use of psychotropic or neuropsychiatric medications.
* A airway assessment with no indication of a difficult intubation including a class I or II Mallampati airway and a mandible-to-hyoid distance of greater than three fingerbreadths.
* Age between 18-75 years.

Exclusion Criteria:

* Does not meet inclusion criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald M Mathews, MD, Principal Investigator — University of Vermont
Locations (1):
- Fletcher Allen Health Care, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No
Data collected was for device algorithm development

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 20 | 20 | 20 | 20
Completed | 19 | 19 | 20 | 17
Not Completed | 1 | 1 | 0 | 3
Not completed — Physician Decision | 1 | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Rocuronium dose 0 mg/kg prior to laryngoscopy
- Group 2: Rocuronium dose 0.2 mg/kg prior to laryngoscopy
- Group 3: Rocuronium dose 0.4 mg/kg prior to laryngoscopy
- Group 4: Rocuronium dose 0.6 mg/kg prior to laryngoscopy
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 19 | 19 | 20 | 17 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (12.3) | 38.6 (14.6) | 39.4 (12.7) | 32.9 (6.4) | 37.9 (11.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 8 | 9 | 34
  Male | 10 | 11 | 12 | 8 | 41

OUTCOME MEASURES:

1. Primary Outcome: The Mean Difference in CVI Between Pre-laryngoscopy and Post-laryngoscopy for Each of the Four Rocuronium Groups
Description: The difference between the mean CVI in three minutes prior to laryngoscopy and three minutes following laryngoscopy reported as the mean change in CVI and the +/- 95% confidence interval for each group.
  The Composite Variability Index (CVI) scale is a logistic regression of three measures of processed electroencephalography (EEG) signals. These signals are Bispectral Index (BIS), the variability of electromyelogram (sEMG), and the variability of BIS (sBIS). The scale ranges from 0 to 100 where a lower CVI value represents a lower likelihood of intraoperative somatic responses, and a higher CVI value represents a higher likelihood of intraoperative somatic responses.
Time Frame: Six minutes after the dose of rocuronium with laryngoscopy at 3 minutes after the study intervention
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Group 1: Rocuronium 0mg/kg
- Group 2: Rocuronium 0.2mg/kg
- Group 3: Rocuronium 0.4mg/kg
- Group 4: Rocuronium 0.6mg/kg
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 20 | 19 | 20 | 16
units on a scale | 2.40 [2.15 to 2.64] | 1.39 [0.95 to 1.83] | 0.48 [0.24 to 0.72] | 0.17 [-0.04 to 0.38]
Statistical Analysis 1: Comparison: Group 1 vs Group 2 vs Group 3 vs Group 4; Null hypothesis that neuromuscular blocking drugs have no effect on CVI with 95% confidence; Test type: Non-Inferiority or Equivalence — Sample size needed for a one-way ANOVA test with an alpha of 0.05 and power of 0.8 to rule out the null hypothesis that neuromuscular blocking drugs have no effect on CVI with 95% confidence was a total of 64 or 16 per Group; p < 0.05, ANOVA — Comparisons of the means were accomplished via student's t-test with Bonferroni correction for multiple comparisons

2. Secondary Outcome: The Average CVI During the Maintenance Phase of Anesthesia for the Two Remifentanil Groups
Description: Mean CVI from incision to propofol off reported as the mean CVI +/- 95% confidence interval for the two groups
Time Frame: Maintenance Anesthesia
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Remifentanil 2ng/ml; Remifentanil 8 ng/ml: The anesthesia provider will titrate propofol as appropriate throughout the procedure to maintain a BIS level between 45- 60.
Arm/Group | Remifentanil 2ng/ml | Remifentanil 8 ng/ml
Number analyzed (Participants) | 33 | 38
units on a scale | 1.73 [1.56 to 1.9] | 1.38 [1.31 to 1.45]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Response to mediations for laryngoscopy in the operating room
Groups:
- Group 1: Rocuronium dose 0 mg/kg
- Group 2: Rocuronium dose 0.2 mg/kg
- Group 3: Rocuronium dose 0.4 mg/kg
- Group 4: Rocuronium dose 0.6 mg/kg
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/20 | 0/17
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/20 | 0/17

LIMITATIONS AND CAVEATS:
Sample size for this study calculation was based upon the assumption that that the expected mean of CVI would be 60 with a variance of 30 and that the variance of 30 would be equal for each group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No